CLINICAL TRIAL: NCT02201771
Title: Compare the Efficacy of Different Antiplatelet Therapy Strategy After Coronary Artery Bypass Graft Surgery
Brief Title: Different Antiplatelet Therapy Strategy After Coronary Artery Bypass Graft Surgery
Acronym: DACAB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Qiang Zhao,MD, Vice President of Ruijin Hospital, Professor and director, Department of Cardiac Surgery, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISSBRIL0211
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Bypass; Antiplatelet Agents
Keywords: CABG; Antiplatelet; Ticagrelor
MeSH Terms: interventions — Aspirin; Ticagrelor

ARMS (3):
- Aspirin (Active Comparator): aspirin 100mg tablet by mouth daily for 12 months
  Interventions: Drug: Aspirin
- Ticagrelor plus Aspirin (Experimental): ticagrelor 90mg tablet by mouth twice daily and aspirin 100mg tablet by mouth daily for 12 months
  Interventions: Drug: Aspirin; Drug: Ticagrelor
- Ticagrelor (Experimental): ticagrelor 90mg tablet by mouth twice daily for 12 months
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Aspirin
  Arms: Aspirin; Ticagrelor plus Aspirin
Drug: Ticagrelor
  Arms: Ticagrelor; Ticagrelor plus Aspirin

SUMMARY:
The study population will include all patients undergoing elective CABG. Consent and randomization will occur before surgery. Total 500 patients undergoing elective CABG will be randomly assigned into three groups with 1:1:1 ratio(167 patients per group) in this open-label study. All the enrolled patients will stop oral antiplatelet drugs according to local protocol before the surgery. Within the first 24 hours after surgery, study medication should be restarted and continued for 12 months. Arm A will restart oral antiplatelet drugs by giving aspirin 100mg qd, Arm B will also restart oral antiplatelet drugs by giving ticagrelor 90mg bid plus aspirin 100mg qd and Arm C will also restart oral antiplatelet drugs by giving ticagrelor 90mg bid. Treatment will continue for 12 months, at which time patients will undergo a multislice computed tomography angiography to assess vein graft patency.

This study is designed to show the superiority of ticagrelor and ticagrelor plus aspirin as compared with aspirin monotherapy respectively for the 1-year primary efficacy end point of vein graft patency.

DETAILED DESCRIPTION:
The study is designed to show the superiority of ticagrelor and ticagrelor plus aspirin as compared with aspirin monotherapy respectively for the 1-year primary efficacy end point of vein graft patency. The primary comparison includes two separate parts. One is to demonstrate T+A better than A and the other is T better than A.

One year rate of vein graft patency in the aspirin group is estimated as 80%. The assumed rate of ticagrelor plus aspirin is 90%. With a two-sided alpha level 0.05 and 80% power, 199 grafts to each group are required. On the other hand, if we assume the rate of ticagrelor monotherapy has the 1-year vein graft patency rate of 87%, under the same two-sided 0.05 alpha 441 grafts in each arm will offer 80% power to show the superiority of ticagrelor along for the primary efficacy end point.

Combined the above two assumptions, if the allocation rate is 1:1:1, this study needs to recruit 1,323 grafts in total (441 in each) to achieve the pre-specified power for both the two comparisons (T+A vs. A and T vs. A).

The principle investigator assumes that the average number of the vien grafts in one patient is 2.7-3.0. With this assumption, 500 patients are to be recruited, which will provide us a total of 1350 - 1500 grafts.

According to the above, this study will be a confirmatory clinical trial to the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to provide written informed consent
* Provision of informed consent prior to any study specific procedures
* Female and male patients aged 18-80 years
* Indication for CABG surgery

Exclusion Criteria:

* Cardiogenic shock, haemodynamic instability
* Need for urgent revascularization within 5 days from presentation
* Single vessel disease
* Two vessel disease with normal left ventricular function (> 50%)
* Need for concomitant other cardiac surgery (e.g. valve replacement)
* Need for dual antiplatelet treatment for the patients undergoing CABG after acute coronary syndrome(ACS)
* Contraindication for aspirin and ticagrelor use(e.g. known allergy)
* History of bleeding diathesis within 3 months prior presentation
* History of significant GI bleed within 1 year prior presentation
* History of peptic ulcer without GI bleeding in past 3 years
* History of intracranial hemorrhage
* History of moderate to severe liver impairment
* Patient requires dialysis
* Patient with an increased risk of bradycardic events (as patients without a pacemaker who have sick sinus syndrome, 2nd or 3rd degree arteriolar-venular block or bradycardic-related syncope)
* Need vitamin K antagonist therapy after bypass surgery eg. persistent atrial fibrillation, mechanical valves
* Known, clinically important thrombocytopenia(i.e. < 100*109/L)
* Known, clinically important anaemia (i.e. <100g/L)
* Participation in another investigational drug or device study in the last 30 days
* Pregnancy or lactation(for premenopausal women 2 methods of reliable contraception, one of which must barrier method, are required)
* Concomitant oral or intravenous therapy with strong cytochrome P450 3A4(CYP3A4) inhibitors, CYP3A4 substrates with narrow therapeutic indices, or strong CYP3A4 inducers which cannot be stopped for the course of the study (strong inhibitors: ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, over 1 litre daily of grapefruit juice. Substrates with narrow therapeutic index: cyclosporine, quinidine. Strong inducers: rifampin, phenytoin, carbamazepine. )
* Any other condition such as active cancer
* Life expectancy less than 12 months that may result in protocol non-compliance or a risk for being lost to follow up
* Indication for major surgery(e.g. cancer treatment, carotid surgery, cerebral surgery, major vascular surgery)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2014-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Zhao, MD.PhD, Principal Investigator — Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, China; Yunpeng Zhu, MD., Study Director — Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, China
Locations (6):
- China (6):
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nan Jing First Hospital, Nanjing, Jiangsu
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Xinhua Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Zhao Q, Zhu Y, Xu Z, Cheng Z, Mei J, Chen X, Wang X. Effect of Ticagrelor Plus Aspirin, Ticagrelor Alone, or Aspirin Alone on Saphenous Vein Graft Patency 1 Year After Coronary Artery Bypass Grafting: A Randomized Clinical Trial. JAMA. 2018 Apr 24;319(16):1677-1686. doi: 10.1001/jama.2018.3197. PMID 29710164

RESULTS

PARTICIPANT FLOW:
Groups:
- Aspirin: aspirin 100mg tablet by mouth daily for 12 months
  Aspirin
- Ticagrelor Plus Aspirin: ticagrelor 90mg tablet by mouth twice daily and aspirin 100mg tablet by mouth daily for 12 months
  Aspirin
  Ticagrelor
- Ticagrelor: ticagrelor 90mg tablet by mouth twice daily for 12 months
  Ticagrelor
Period: Overall Study
Arm/Group | Aspirin | Ticagrelor Plus Aspirin | Ticagrelor
Started | 166 | 168 | 166
Completed | 153 | 158 | 156
Not Completed | 13 | 10 | 10
Not completed — Death | 3 | 2 | 0
Not completed — Protocol Violation | 10 | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin | Ticagrelor Plus Aspirin | Ticagrelor | Total
Number analyzed (Participants) | 166 | 168 | 166 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (8.1) | 63.5 (8.2) | 63.3 (8.3) | 63.6 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 34 | 32 | 91
  Male | 141 | 134 | 134 | 409
Region of Enrollment [Number; unit: participants]
  China | 166 | 168 | 166 | 500

OUTCOME MEASURES:

1. Primary Outcome: The Patency of Saphenous Vein Grafts
Description: assessed by multislice computed tomography angiography (MSCTA) or coronary angiography(CAG). FitzGibbon grade A (stenosis <50%) is defined as "patency".
Time Frame: up to 12 months
Population: ITT analysis, Patients with missing data were considered to have occluded saphenous vein grafts.
Measure: Number (95% Confidence Interval); unit: percentage of patent SV grafts
Units Other Than Participants: saphenous vein grafts
Arm/Group | Aspirin | Ticagrelor Plus Aspirin | Ticagrelor
Number analyzed (Participants) | 166 | 168 | 166
Number analyzed (saphenous vein grafts) | 485 | 487 | 488
percentage of patent SV grafts | 76.5 [70.8 to 82.1] | 88.7 [84.6 to 92.8] | 82.8 [78.0 to 87.6]

2. Secondary Outcome: The Patency of Saphenous Vein Grafts
Description: assessed by MSCTA or CAG. FitzGibbon grade A (stenosis <50%) is defined as "patency".
Time Frame: up to 7 days
Measure: Number (95% Confidence Interval); unit: percentage of patent SV grafts
Units Other Than Participants: saphenous vein grafts
Arm/Group | Aspirin | Ticagrelor Plus Aspirin | Ticagrelor
Number analyzed (Participants) | 166 | 168 | 166
Number analyzed (saphenous vein grafts) | 485 | 487 | 488
percentage of patent SV grafts | 91.1 [87.4 to 94.8] | 94.9 [92.2 to 97.6] | 94.3 [91.8 to 96.7]

3. Secondary Outcome: The Rate of Post-operative Atrial Fibrillation After CABG.
Description: Number of Participants with Post-operative Atrial Fibrillation after CABG
Time Frame: up to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Ticagrelor Plus Aspirin | Ticagrelor
Number analyzed (Participants) | 166 | 168 | 166
Participants | 23 | 20 | 13

4. Secondary Outcome: The Rate of Freedom From Angina According to Canadian Cardiovascular Society (CCS) Classification
Description: Number of Participants Free of Angina per CCS Classification
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Ticagrelor Plus Aspirin | Ticagrelor
Number analyzed (Participants) | 166 | 168 | 166
Participants | 154 | 158 | 155

5. Secondary Outcome: The Number of Major Adverse Cardiovascular Event (MACE)
Description: MACE, composite of CV death, myocardial infarction or stroke (ischaemic or unknown etiology)
Time Frame: up to 12 months
Measure: Number; unit: events
Arm/Group | Aspirin | Ticagrelor Plus Aspirin | Ticagrelor
Number analyzed (Participants) | 166 | 168 | 166
events | 9 | 4 | 3

6. Secondary Outcome: Number of the Major Bleeding Events
Description: According to modified TIMI criteria, the "Major Bleeding Events" is defined as the combination of CABG-related bleeding and non-CABG-related major bleeding(Intracranial bleeding, Clinically overt signs of hemorrhage with hemoglobin drop ≥5 g/dL and Fatal bleeding).
Time Frame: up to 12 months
Measure: Number; unit: events
Arm/Group | Aspirin | Ticagrelor Plus Aspirin | Ticagrelor
Number analyzed (Participants) | 166 | 168 | 166
events | 0 | 3 | 2

7. Other Pre Specified Outcome: The Rate of Gastroduodenal Injury Assessed by Esophagogastroduodenoscopy (EGD)
Description: Not all but the patients recruited in Ruijin Hospital
Time Frame: at 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Aspirin | Ticagrelor Plus Aspirin | Ticagrelor
All-Cause Mortality (participants affected / at risk) | 3/166 | 2/168 | 0/166
Serious Adverse Events (participants affected / at risk) | 9/166 | 3/168 | 3/166
Other Adverse Events (participants affected / at risk) | 78/166 | 91/168 | 74/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aspirin (N=166) | Ticagrelor Plus Aspirin (N=168) | Ticagrelor (N=166)
Nonfatal myocardial infarction (Cardiac disorders) | 3 | 2 | 2
Nonfatal stroke (Cardiac disorders) | 4 | 0 | 2
Cardiovascular death (Cardiac disorders) | 2 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aspirin (N=166) | Ticagrelor Plus Aspirin (N=168) | Ticagrelor (N=166)
Atrial Fibrillation (Cardiac disorders) | 25 | 22 | 15
Perioperative myocardial injury (Cardiac disorders) | 11 | 25 | 14 — cTn > 10*URL but not myocardial infarction
Hypoproteinemia (Metabolism and nutrition disorders) | 17 | 22 | 18 — serum albumin<25g/L
Anaemia (Blood and lymphatic system disorders) | 14 | 10 | 12 — Hemoglobin < 70g/L
Renal disfunction (Renal and urinary disorders) | 6 | 12 | 9 — Serum creatinine>200umol/L
Incision complication (Injury, poisoning and procedural complications) | 10 | 9 | 6 — poor healing of incision

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT02201771/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT02201771/SAP_001.pdf